CLINICAL TRIAL: NCT04326608
Title: Psycho-social Aspects After a Physiotherapy Intervention in Chronic TMD Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Gema Serrano-Hernanz, PhD, Universidad Complutense de Madrid
Other Study IDs: Geserrher
Record Dates: First submitted 2020-03-19; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: TMD
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: physiotherapy — manual therapy and sef-care exercises

SUMMARY:
How patients psycho-social factors change after a physical intervention in patients with chronic TMD pain

ELIGIBILITY:
Inclusion Criteria:

* Chronic myofascial TMD pain

Exclusion Criteria:

* Neurologic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic TMD pain
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
TSK-11 | immediately after treatment
  Tampa Scale for Kinesiophobia
TSK-11 | at 3 months
  Tampa Scale for Kinesiophobia

IPD SHARING:
Plan to Share IPD: No